CLINICAL TRIAL: NCT01463774
Title: Pivotal BE CANA/MET IR FDC - Low Strength
Brief Title: A Study to Assess the Bioequivalence of 2 Fixed Dose Combination Tablets of Canagliflozin and Metformin Immediate Release (IR) With Respect to the Individual Components of Canagliflozin and Metformin IR Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100674; 28431754DIA1039 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-09-20; First posted 2011-11-02 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Bioequivalence; Canagliflozin (JNJ-28431754); Metformin
MeSH Terms: interventions — Metformin

ARMS (2):
- Treatment Sequence AB (Experimental): The study consists of 2 treatment periods (A and B). Each treatment period wiill be separated by a washout period of 10-15 days.
  Interventions: Drug: Treatment A: Canagliflozin tablet; Drug: Treatment A: Metformin IR tablets; Drug: Treatment B: Canagliflozin/metformin fixed dose combination tablets
- Treatment Sequence BA (Experimental): The study consists of 2 treatment periods (A and B). Each treatment period wiill be separated by a washout period of 10-15 days.
  Interventions: Drug: Treatment A: Canagliflozin tablet; Drug: Treatment A: Metformin IR tablets; Drug: Treatment B: Canagliflozin/metformin fixed dose combination tablets

INTERVENTIONS:
Drug: Treatment A: Canagliflozin tablet — Type=exact number, unit=mg, number=100, form=tablet, route=oral use. One canagliflozin tablet taken orally (by mouth) on Day 1 of Treatment Period A.
Drug: Treatment A: Metformin IR tablets — Type=exact number, unit=mg, number=850, form=tablet, route=oral use. Two metformin IR tablets taken orally (by mouth) on Day 1 of Treatment Period A.
Drug: Treatment B: Canagliflozin/metformin fixed dose combination tablets — Type=exact number, unit=mg, number=50/850, form=tablet, route=oral use. Two canagliflozin/metformin IR tablets taken orally (by mouth) on Day 1 of Treatment Period B.

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of a fixed dose combination tablet of canagliflozin and metformin immediate release (IR) in comparison with the individual components of canagliflozin and metformin IR.

DETAILED DESCRIPTION:
This is an open-label (identity of study drug will be known to volunteer and study staff), single-center study to evaluate the bioequivalence of canagliflozin and metformin when administered orally (by mouth) as individual components (ie, separate tablets of canagliflozin and metformin) (Treatment A) and when administered as a fixed dose combination tablet (ie, canagliflozin and metformin in the same tablet) (Treatment B). Healthy volunteers participating in the study will be randomly (by chance) assigned to receive Treatment A followed by Treatment B or Treatment B followed by Treatment A with a period of approximately 15 days between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 30 kg/m² inclusive and a body weight of not less than 50 kg

Exclusion Criteria:

* History of or current medical illness, abnormal values for hematology or clinical chemistry laboratory tests, or abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) deemed to be clinically significant by the Investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Canagliflozin plasma concentrations | Up to 72 hours
Metformin plasma concentrations | Up to 72 hours

SECONDARY OUTCOMES:
Adverse events | Up to approxmately 23 days
  The number and type of adverse events will be reported from Day 1 of treatment period 1 through 7-10 days after treatment period 2 including the 10-15 washout period between treatment periods (total time is approximately 23 days).
Changes from baseline in clinical laboratory test results | Up to approximately 23 days
Vital Signs | Up to approximately 23 days
  Blood pressure, pulse, and oral body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC L.LC. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Lincoln, Nebraska, United States